CLINICAL TRIAL: NCT02947763
Title: Healing Rates After Single Versus Multiple Visits Endodontic Treatment of Necrotic Teeth With Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Single Versus Multiple Visits Endodontic Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Safeya AbdelRahaman Hassan, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-10-231
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Periapical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Ciprofloxacin; Minocycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- multiple visit (Active Comparator): multiple visit root canal treatment with triple antibiotic paste intracanal medication (a mixture of metronidazole, ciprofloxacin, and minocycline)
  Interventions: Drug: mixture of metronidazole, ciprofloxacin, and minocycline
- single visit (No Intervention): single visit root canal treatment without any intra-canal medication

INTERVENTIONS:
Drug: mixture of metronidazole, ciprofloxacin, and minocycline — placement of intracanal medication
  Other Names: no other names
  Arms: multiple visit

SUMMARY:
Healing rate after single visit or multiple visit endodontic treatment using triple paste intracanal medicament will be assessed both clinically and radio-graphically for follow-up period up to one year

DETAILED DESCRIPTION:
Patients with necrotic teeth with apical periodontitis will be selected according to the eligibility criteria and patients are then randomized to either single visit or multiple visit using triple paste intracanal medicament. Postoperative pain will then assessed using numerical rating scale after 1, 2, 3 and 7 days post-instrumentation. Radiographic healing will be assessed every 3 months up to one year.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients; age between 16-55 years old.
2. Males or Females.
3. Maxillary or mandibular single-root tooth or a multi-rooted tooth with:

   * Non-vital response of pulp tissue.
   * Radiographic evidence of periapical lesions (minimum size 2.0 mm × 2.0 mm) related to one root in case of multi-rooted teeth.
   * Asymptomatic patients.
4. Positive patients' acceptance for participation in the study.

Exclusion Criteria:

1. Primary teeth, and permanent teeth with immature apex.
2. Teeth previously accessed or endodontically treated.
3. Patients with diabetes and immune-compromising disease.
4. Patients allergic to metronidazole, ciprofloxacin, or minocycline.
5. Vital cases or necrotic without periapical lesion.
6. Pregnant women.
7. Teeth with unfavorable conditions for rubber-dam application.
8. Tooth associated with vertical root fracture, coronal perforation, calcification and external or internal root resorption.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 24 hours
  using numerical rating scale from 0-10
postoperative pain | 48 hours
  using numerical rating scale from 0-10
postoperative pain | 72 hours
  using numerical rating scale from 0-10
postoperative pain | 7 days
  using numerical rating scale from 0-10

SECONDARY OUTCOMES:
Radiographic healing | 3 months
  using digital radiography
Radiographic healing | 6 months
  using digital radiography
Radiographic healing | 9 months
  using digital radiography
Radiographic healing | 12 months
  using digital radiography

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] AbdurRahman S, Abdel Aziz SM, Gawdat SI, AbdalSamad AM. Postoperative pain of patients with necrotic teeth with apical periodontitis following single visit endodontic treatment versus multiple visit endodontic treatment using triple antibiotic paste: a randomized clinical trial. F1000Res. 2019 Jul 26;8:1203. doi: 10.12688/f1000research.19936.1. eCollection 2019. PMID 32047601